CLINICAL TRIAL: NCT02001571
Title: A Phase 1 Single Dose Open-Label Pharmacokinetic Study of Abiraterone Acetate in Male Participants With Mild or Moderate Hepatic Impairment Compared to Matched Control Participants With Normal Hepatic Function
Brief Title: A Study to Assess the Effect of Abiraterone Acetate in Male Participants With Mild or Moderate Hepatic Impairment Compared to Matched Control Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016948; COU-AA-011 (Other: Cougar Biotechnology, Inc.)
Record Dates: First submitted 2013-10-31; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Abiraterone acetate; Pharmacokinetics
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Mild Hepatic participants administered to four 250 mg tablets (1000 mg) orally on Day 1.
  Interventions: Drug: Abiraterone acetate
- Cohort 2 (Experimental): Moderate Hepatic participants administered to four 250 mg tablets (1000 mg) orally on Day 1.
  Interventions: Drug: Abiraterone acetate
- Cohort 3 (Experimental): Normal Hepatic participants administered to four 250 mg tablets (1000 mg) orally on Day 1.
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Abiraterone acetate — On the morning of Day 1, each participant was given four 250 mg tablets of abiraterone acetate with 240 mL of room temperature tap water. Dosing followed at least a 10-hour fast from food (not including water).

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (study of what the body does to a drug) of 1000 mg oral dose of abiraterone acetate and its major metabolite(s) with mild or moderate hepatic impairment and matched control Participants with normal hepatic function.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) pharmacokinetics and safety study of abiraterone acetate administered as four 250 mg tablets (1000 mg) to 3 cohorts (groups) in Cohort 1 (Mild Hepatic Impairment), Cohort 2 (Moderate Hepatic Impairment) and Cohort 3 (Normal Hepatic Function). There will be approximately 8 Participants per cohort (total of approximately 24 Participants for the study). The cohorts will be dosed sequentially and activities will consist of Screening, Study and Follow-up periods, a total of up to approximately 36 days. Possible Participants will be screened to assess their eligibility to enter the study within 14 days prior to study Day 1. Participants will be confined at the Clinical Research Center (CRC) from the time of Check-in on Day -1 until discharge on Day 5. Participants will return to the CRC on Days 8 and 15 and there will be a follow-up call or visit on Day 22. A review of all clinical and laboratory data through Day 8 evaluations in each cohort will be done by the Medical Monitor and the Principal Investigator (PI) prior to proceeding with dosing any further cohort, if indicated. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Non smokers or light smokers and willing to limit smoking for the period of confinement to 4 cigarettes per day
* Body Mass Index of 18-35 kg/m2
* Negative test for breathalyzer alcohol and drugs of abuse and HIV antibody test at Screening
* Agrees to protocol-defined use of effective contraception
* Participants with Mild or Moderate Hepatic Impairment
* Must have mild or moderate hepatic impairment
* On a stable dose of medication and/or treatment regimen for at least 2 weeks before dosing as well as during the study
* Clinical laboratory evaluations within the reference range for the test laboratory
* Participants with normal hepatic function have no clinically significant findings from medical history, physical examination, Laboratory values within protocol defined parameters

Exclusion Criteria:

* Any other investigational study drug trial within 5 half-lives of that investigational study drug or 30 days prior to dosing with Abiraterone acetate, whichever is longer
* Inability to swallow four (4) 250 mg abiraterone acetate tablets
* History of or current clinically significant medical illness that would potentially alter absorption and/or excretion of orally administered drugs
* History or presence of a clinically significant abnormal ECG
* Donation of blood or significant loss of blood within 56 days prior to Day 1 or planned donation of blood or plasma from Screening through 30 days after Day 1
* Use of any prescription medications/products or any OTC, non-prescription unrelated to existing allowable stable medical conditions within 5 half-lives of that product or 7 days prior to dosing with abiraterone acetate, whichever is longer
* Clinically significant renal laboratory findings
* Participants with Mild or Moderate Hepatic Impairment will be excluded - any significant medical history other than hepatic impairment that may affect the interpretation of the data or which otherwise contraindicates participation in the study
* Acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within 2 weeks
* Autoimmune liver disease; Esophageal variceal bleeding within 6 months prior to Screening, unless successfully treated with banding, Gastric varices
* Spontaneous bacterial peritonitis within 3 months prior to Screening
* Portosystemic shunt, Organ transplant, Wilson's disease, Cholestatic liver disease (e g , primary biliary cirrhosis or primary sclerosing cholangitis)
* Clinically significant laboratory findings except as related to hepatic impairment
* Control Participants with Normal Hepatic Function Any significant laboratory results, including specifically Positive for Hepatitis B or C, Hemoglobin < 12 0 g/dL LFTs outside of normal limits

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of abiraterone acetate | Up to 96 hours postdose

SECONDARY OUTCOMES:
The number of Participants with adverse events | Approximately 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (1):
- Orlando, Florida, United States

REFERENCES:
- [Derived] Marbury T, Lawitz E, Stonerock R, Gonzalez M, Jiao J, Breeding J, Haqq C, Verboven P, Stieltjes H, Yu M, Molina A, Acharya M, Chien C, Tran N. Single-dose pharmacokinetic studies of abiraterone acetate in men with hepatic or renal impairment. J Clin Pharmacol. 2014 Jul;54(7):732-41. doi: 10.1002/jcph.253. Epub 2014 Jan 17. PMID 24374856